CLINICAL TRIAL: NCT01486251
Title: Assessment of the Tumor Vascular Effects of the Pan-vegfr Tyrosine Kinase Inhibitor Axitinib Using Dynamic Contrast-enhanced Ultrasonography (Dce-us) in Patients With Refractory Metastatic Colorectal Cancer
Brief Title: Assessment of Tumor Vascular Effects of Axitinib With Dynamic Ultrasonography in Patients With Metastatic Colorectal Cancer
Acronym: AXUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011-001151-37; 2011/1738 (Other: CSET number)
Record Dates: First submitted 2011-10-31; First posted 2011-12-06 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental (Experimental): axitinib will be given BID orally. One cycle is defined as a 14-day period (7 days ON / 7 days OFF). The 3 dose levels tested will be: 1st cycle: 5 mg BID; 2nd cycle: 7 mg BID; 3rd cycle: 10 mg BID.
  Patients will receive a first cycle of single agent axitinib at the starting dose with DCE-US assessment. If no study treatment-related adverse event (AE) of grade > 1 is observed during this cycle, intrapatient dose escalation will be performed for the second cycle. The same dose escalation method wil apply between the 2d and 3d cycles.
  Interventions: Drug: axitinib

INTERVENTIONS:
Drug: axitinib — Axitinib will be given BID orally. The 3 dose levels tested will be: 1st cycle: 5 mg BID; 2nd cycle: 7 mg BID; 3rd cycle: 10 mg BID.
  One cycle is defined as a 14-day period (7 days ON / 7 days OFF). Patients will receive a first cycle of single agent axitinib at the starting dose with DCE-US assessment. If no study treatment-related adverse event (AE) of grade > 1 is observed during this cycle, intrapatient dose escalation will be performed for the second cycle. The same dose escalation method wil apply between the 2d and 3d cycles.

SUMMARY:
The purpose of this study is to evaluate and quantify the dynamic modifications of tumor blood perfusion on axitinib therapy in patients with refractory mCRC for each dose of Axitinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of CRC
* Measurable metastatic disease to the liver in proven disease progression (according to RECIST criteria) at baseline (within 4 weeks prior to study entry), with at least one lesion > 2cm considered appropriate for DCE-US examination
* Previously exposed to at least, irinotecan, oxaliplatin and a fluoropyrimidine, all 3 administered at optimal doses, over one or two chemotherapy (CT) lines for metastatic disease with a clear resistance to these drugs. Previous exposure to bevacizumab and/or anti-EGFR monoclonal antibody is allowed.
* Age ≥18 years; Performance Status (PS) 0-2 and life expectancy > 3 months.
* Adequate biological functions: Neutrophils ≥ 1.5 x 109/L; Platelets ≥ 100 x 109/L; Hemoglobin > 9 g/dl; Creatinine clearance > 30 ml/min (cockcroft & Gault formula). Serum bilirubin < 1,5 x the upper normal limit (UNL) and AST/ALT < 5 x UNL.
* Signed written informed consent
* Female patients with childbearing potential (<2 years after last menstruation) and male must use effective means of contraception during the study treatment and at least 6 months after the last study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Echography measure | baseline and on day 2, day 7, day 15, day 29, day 35 and day 43
  Variation of the total area under the curve (tAUC) measured by DCE-US in the region of interest (ROI) between baseline and the end of each axitinib cycle at increasing dose.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ducreux, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut gustave roussy, Villejuif, France